CLINICAL TRIAL: NCT03902158
Title: Use of Virtual Reality Glasses as an Audiovisual Distraction Technique During Anesthesia in Behavior, Anxiety and Pain Perception in Children
Brief Title: Use of Virtual Reality Glasses During Anesthesia in Behavior, Anxiety and Pain Perception of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Clinical Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PPGO 0028
Record Dates: First submitted 2019-01-22; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glasses (Experimental)
  Interventions: Device: Glasses; Behavioral: Distraction techniques
- Distraction techniques (No Intervention): No glasses will be used

INTERVENTIONS:
Device: Glasses — The patient will wear virtual reality glasses during anesthesia
  Arms: Glasses
Behavioral: Distraction techniques — The patient will undergo distraction techniques
  Arms: Glasses

SUMMARY:
One of the most challenging aspects of Pediatric Dentistry is the management of child behavior. Among the procedures performed, local anesthesia is one of the factors that influence the increase in fear and anxiety in children in relation to dental procedures. This study aims to evaluate the effect of the use of virtual reality glasses as an audiovisual distraction technique during anesthesia in behavior, anxiety and pain perception, comparing it with traditional behavior management techniques. A sample of 44 children was estimated and will be selected with the following inclusion criteria: be between 5 and 9 years of age; good general health; no prior dental experience involving anesthesia in the last 2 years; need for restorative treatment or exodontia under local anesthesia. Children with physical or mental disabilities will be excluded and those who report poor behavior in dental consultations will be excluded. The sample will be randomized with 22 envelopes for the group that will use the glasses during the procedure(G0) and 22 envelopes containing group that will not use the glasses in consultation (G1).

The treatments will be performed in 2 visits, the first for initial examination, and the other for performing the procedures are either extraction or restorative treatment with the use of local anesthesia. During dental treatment, the dentist will explain the procedure in layman's terms using the basic techniques of behavior management, such as the "tell-show-do" technique, positive reinforcement, conventional distraction in all consultations. When using the distraction technique with virtual reality during the procedure, the virtual stereo glasses model HDMI-MHL 98 Inches (98') will be used. In all two consultations, VENHAM anxiety will be assessed through VENHAM scale and heart rate measurement at the beginning, during and at the end of the visit, as well as the perception of pain during the procedure (FLACC) and after finishing the service through the FPS-R scale. During the visits, the data will be collected using a previously tested tab. The data will be entered into a worksheet in the Microsoft® Excel® 2016 program and analyzed in the Stata 14.0 program. There will be a single blind blinding: both for the typist and who will analyze the data. A descriptive analysis of the data will be performed, obtaining the absolute and relative frequencies. Comparisons in the outcomes of interest between groups G0 and G1 will be performed using the chi-square test for dichotomous variables and the t-test for comparison of means. A significance level of 5% will be adopted for all analyzes.

DETAILED DESCRIPTION:
One of the most challenging aspects of Pediatric Dentistry is the management of child behavior. Anxiety is often manifested by children during dental appointments, and may represent a challenge in the dental surgeon's clinical practice. Among the procedures performed, local anesthesia is one of the factors that influence the increase in fear and anxiety in children in relation to dental procedures. In view of the basic techniques used to manage children's behavior, distraction has been widely used to provide a more relaxed and effective experience during dental treatment for children. Thus, this study aims to evaluate the effect of the use of virtual reality glasses as an audiovisual distraction technique during anesthesia in behavior, anxiety and pain perception, comparing it with traditional behavior management techniques. A sample of 44 children was estimated and will be selected with the following inclusion criteria: be between 5 and 9 years of age; good general health; no prior dental experience involving anesthesia in the last 2 years; need for restorative treatment or exodontia under local anesthesia. Children with physical or mental disabilities will be excluded and those who report poor behavior in dental consultations will be excluded. The sample will be randomized through the draw of envelopes at the time of the service, being 22 envelopes for the group that will use the glasses during the procedure(G0) and 22 envelopes containing group that will not use the glasses in consultation (G1).

The treatments will be performed in 2 visits, the first for initial examination, and the other for performing the procedures are either extraction or restorative treatment with the use of local anesthesia. During dental treatment, the dentist will explain the procedure in layman's terms using the basic techniques of behavior management, such as the "tell-show-do" technique, positive reinforcement, conventional distraction in all consultations. When using the distraction technique with virtual reality during the procedure, the virtual stereo glasses model HDMI-MHL 98 Inches (98) will be used. In all two consultations, VENHAM anxiety will be assessed through VENHAM scale and heart rate measurement at the beginning, during and at the end of the visit, as well as the perception of pain during the procedure (FLACC) and after finishing the service through the FPS-R scale. During the visits, the data will be collected using a previously tested tab. The data will be entered into a worksheet in the Microsoft® Excel® 2016 program and analyzed in the Stata 14.0 program. There will be a single blind blinding: both for the typist and who will analyze the data. A descriptive analysis of the data will be performed, obtaining the absolute and relative frequencies. Comparisons in the outcomes of interest between groups G0 and G1 will be performed using the chi-square test for dichotomous variables and the t-test for comparison of means. A significance level of 5% will be adopted for all analyzes.

ELIGIBILITY:
Inclusion Criteria:

* good general health;
* no prior dental experience involving anesthesia in the last 2 years;
* need for restorative treatment or exodontia under local anesthesia.

Exclusion Criteria:

* physical or mental disabilities;
* report of poor behavior during dental treatment.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Perception of pain | 5 minutes after anesthesia, i.e., after anesthesia, VAS will be performed in a maximum of 5 minutes after anesthesia
  Visual analogue scale (VAS) will be used to measure pain immediately after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Pelotas, Rio Grande do Sul, Brazil